CLINICAL TRIAL: NCT03697551
Title: A Non-Randomised Phase II Study to Evaluate the Optimal Uptake Time of 68GA-OPS202 as a sstr2 Positive PET Imaging Agent in Subjects With Newly Diagnosed Breast Cancer
Brief Title: Define the Optimal Uptake Time of 68Ga-OPS202 When Used as a PET (Positron Emission Tomography) Imaging Agent in Subjects With Newly Diagnosed Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment challenges and not due to safety concerns.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D-FR-01070-003; 2018-000028-33 (EudraCT Number)
Record Dates: First submitted 2018-07-12; First posted 2018-10-05 (Actual); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-OPS202 (Experimental): A single dose of Satoreotide trizoxetan will be administered as a slow intravenous (i.v.) bolus injected over 1 minute at Baseline/Day 1.
  Interventions: Drug: Satoreotide trizoxetan

INTERVENTIONS:
Drug: Satoreotide trizoxetan — Subjects will receive a single dose of Satoreotide trizoxetan consisting of a peptide mass up to 45 μg, with a radioactivity range of 150-200 MBq. Satoreotide trizoxetan is intended for diagnostic use as a Positron emission tomography/computed tomography (PET/CT) tracer for the imaging of tumours expressing SSTR2.
  Other Names: 68Ga-OPS202; 68Ga-IPN01070

SUMMARY:
The purpose of this clinical research is to define the optimal uptake time of 68Ga-OPS202 as a PET imaging agent to be used to detect and localize breast cancer somatostatin receptor subtype 2 (SSTR2) positive lesions.

68Ga-OPS202 is a radiolabelled imaging agent to be used in association with PET. 68Ga-OPS202 is made of two main components: 1) OPS202, an antagonistic somatostatin analogue which binds to the somatostatin receptor (type 2) present on the surface of the tumor cells and 2) Gallium 68, a radioisotope that, combined with OPS202, can be seen in the PET scanner.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older
* Subjects with newly diagnosed (early or advanced) breast cancer
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Adequate bone marrow, liver and renal function, with:

  * Calculated glomerular filtration rate (GFR): ≥45 mL/min
  * Albumin: >30 g/L
  * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (AP): ≤5 times upper limit of normal (ULN)
  * Bilirubin: ≤3xULN (3×1.1 mg/dL)
  * Leukocytes: ≥3x109/L, and neutrophils: ≥1x109/L
  * Erythrocytes: ≥3.5x1012/L
  * Platelets: ≥90x109/L
* Signed written informed consent prior to any study-related procedures.

Exclusion Criteria:

* Subject with resected primary tumour
* Subjects with confirmed ductal carcinoma in situ
* Men with breast cancer
* Presence of an active infection at screening or history of a serious infection within the previous 6 weeks prior to the first 68Ga-OPS202 administration that might interfere with the PET and/or CT analysis
* Subjects who have received any therapy for breast cancer
* Prior or planned administration of a radiopharmaceutical within 8 half-lives of the radionuclide
* Clinically relevant trauma within 2 weeks prior to first 68Ga-OPS202 administration
* Any condition that precludes the proper performance of PET and/or CT scan:

  * Subjects who are not able to tolerate the CT contrast agent
  * Subjects with metal implants or arthroplasty, or any other objects that might interfere with the PET and/or CT analysis
  * Subjects unable to raise arms for prolonged imaging purposes
  * Subjects unable to lie still for the entire imaging time
  * Subjects weighing greater than 110 kg (243 lb)
* Known hypersensitivity to radiolabelled NODAGA (1,4,7- triazacyclononane,1-glutaric acid 4,7 acetic acid), to Gallium-68, to somatostatin analogue peptide JR11 or to any of the excipients of 68Ga- OPS202
* History of, or current active allergic or autoimmune disease, including asthma or any condition requiring long-term use of systemic corticosteroids
* Known human immunodeficiency virus (HIV) or positive serology for HIV, hepatitis B or C
* Administration of another investigational medicinal product within 30 days prior to first 68Ga-OPS202 administration
* Subjects who are pregnant, breast feeding or of childbearing potential not willing to practice effective contraceptive techniques during the study treatment period and for 30 days after the last dose of 68Ga-OPS202 administration; pregnancy test must be performed at the start of the study and prior to 68Ga-OPS202 administration
* Subjects who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study, including any mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study, and/or evidence of an uncooperative attitude
* Subject who experienced a previous cancer (except basocellular carcinoma of the skin and/or in situ carcinoma of the cervix/uterus), and/or subjects treated with curative intent and free from disease for more than 5 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Medical University Innsbruck, Innsbruck, Austria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Female subjects with newly diagnosed breast cancer who had a somatostatin receptor subtype 2 (sstr2) positive lesion were recruited to this study from 22 October 2018, and the last subject last visit was on 6 February 2019. The study was terminated early on 9 August 2019.
Pre-assignment Details: Six subjects were screened and 4 subjects were eligible to receive gallium-68 (68Ga)-satoreotide trizoxetan (formerly 68Ga-OPS202) as a sstr2 positive positron emission tomography (PET) imaging agent. The screening period was up to 14 days prior to the 68Ga-satoreotide trizoxetan administration on Day 1, with a follow-up visit at Day 14.
Groups:
- 68Ga-Satoreotide Trizoxetan: A single dose of 68Ga-satoreotide trizoxetan was administered as a slow intravenous (iv) bolus injected over 1 minute on Day 1.
  The planned, per protocol single dose of 68Ga-satoreotide trizoxetan consisted of a peptide mass up to 45 micrograms, with a radioactivity range of 150-200 megabecquerel (MBq).
Period: Overall Study
Arm/Group | 68Ga-Satoreotide Trizoxetan
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 68Ga-Satoreotide Trizoxetan: A single dose of 68Ga-satoreotide trizoxetan was administered as a slow iv bolus injected over 1 minute on Day 1.
  The planned, per protocol single dose of 68Ga-satoreotide trizoxetan consisted of a peptide mass up to 45 micrograms, with a radioactivity range of 150-200 MBq.
Arm/Group | 68Ga-Satoreotide Trizoxetan
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Sufficiently Avid Lesion(s) Identified as a sstr2 Positive Lesion (Co-Primary Endpoint)
Description: The percentage of subjects with sufficiently avid lesion(s) to be identified as a sstr2 positive lesion using 68Ga-satoreotide trizoxetan was to be determined.
Time Frame: At 0.5, 1.0 and 2.0 hours post injection on Day 1.
Population: The study was stopped prematurely and only four patients were imaged, of whom only three evaluable. No summary statistics are available given the limited data from the small number of evaluable patients and individual patient data are also not presented to protect the privacy of the individuals.
Arm/Group | 68Ga-Satoreotide Trizoxetan
Number analyzed (Participants) | 0

2. Primary Outcome: Differences in the Number of Lesions Detected by 68Ga-Satoreotide Trizoxetan Between the 3 PET Acquisition Timepoints in Primary Breast Lesions (Co-Primary Endpoint)
Description: The differences in the number of lesions detected by 68Ga-satoreotide trizoxetan between the 3 PET acquisition timepoints, and reader interpretation was to be determined.
Time Frame: 0.5, 1.0 and 2.0 hours post injection on Day 1
Population: as for outcome 1
Arm/Group | 68Ga-Satoreotide Trizoxetan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were monitored from Day 1 up to Day 14 (+/- 3 days) (2 weeks).
Arm/Group | 68Ga-Satoreotide Trizoxetan
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
The study was terminated early on 9 August 2019 due to recruitment challenges and the potential overlap with another Ipsen study, and not due to safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT03697551/SAP_000.pdf
  • Study Protocol (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT03697551/Prot_001.pdf